CLINICAL TRIAL: NCT04495751
Title: FOCUS - Pilot Study of Muscadine Grape Extract to Improve Fatigue Among Older Adult Cancer Survivors
Brief Title: Muscadine Grape Extract to Improve Fatigue
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00067614; WFBCCC 98320 (Other: Wake Forest Baptist Comprehensive Cancer Center); UL1TR001420 (NIH); P30CA012197 (NIH)
Record Dates: First submitted 2020-07-28; First posted 2020-08-03 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Fatigue
Keywords: Older; Cancer; Survivors
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double blind study. Only the investigational pharmacists and the statisticians will be unblinded. The blind will be maintained until the study is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Muscadine Grape Extract Arm (Experimental): Muscadine grape extract pill (12 week supply)
  Interventions: Dietary Supplement: Muscadine grape extract; Other: Quality of Life Assessment; Other: Questionnaires; Other: Participant Feedback
- Placebo Arm (Placebo Comparator): Placebo provided (12 week supply)
  Interventions: Drug: Placebo; Other: Quality of Life Assessment; Other: Questionnaires; Other: Participant Feedback

INTERVENTIONS:
Dietary Supplement: Muscadine grape extract — Four pills twice daily
  Arms: Muscadine Grape Extract Arm
Drug: Placebo — Four pills twice daily.
  Arms: Placebo Arm
Other: Quality of Life Assessment — Ancillary studies
Other: Questionnaires — Ancillary studies
Other: Participant Feedback — Ancillary studies

SUMMARY:
The purpose of this research is to see if muscadine grape extract improves fatigue in people age 70 and above who have a history of treated cancer and report the symptom of fatigue.

DETAILED DESCRIPTION:
Primary Objective: To evaluate whether administration of MGE supplementation decreases PROMIS Fatigue score from baseline to 12 weeks compared to placebo.

Secondary Objective(s)

* To evaluate whether administration of muscadine grape extract supplementation (4 tablets twice daily) causes changes in physical function (Pepper Assessment Tool for Disability [PAT-D], Short Physical Performance Battery), physical fitness (6-minute walk), physical activity (Minnesota Leisure Questionnaire), sedentary behavior (Sedentary Behavior Questionnaire) from baseline to 12 weeks compared to placebo.
* To compare changes in health related quality of life (PROMIS Global Health) at 12 weeks in participants randomized to muscadine grape extract group vs. placebo.
* To compare changes in the Fried frailty index at 12 weeks in participants randomized to muscadine grape extract vs. placebo.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive muscadine grape extract orally (PO) twice daily (BID) for 12 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO BID for 12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study, patients are followed up for 30 days after the last dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported history of cancer diagnosed > 12 months prior to enrollment excluding non-melanoma skin cancer with no evidence of disease at enrollment.
* Eligible solid tumor cancer types include Stage 1-3 breast, lung, head and neck, colorectal, anal, prostate, melanoma, bladder/ureteral, esophageal, gastric, pancreatic, kidney, liver/biliary, uterine, cervical, ovarian, sarcoma. (superficial disease and in situ disease only is excluded)
* Eligible hematologic malignancies include lymphoma any subtype any stage in remission, multiple myeloma in remission, leukemia any subtype in remission.
* Eligible prior cancer treatment modalities include surgery, radiation, chemotherapy, hormonal therapies, immunotherapy, biologic therapies.
* All anti-cancer therapy completed > 12 months prior to enrollment
* Age 65 years and older
* Presence of self-reported fatigue defined by a response of "somewhat, quite a bit or very much" to the screening question "During the past seven days, did you feel fatigued: Not at all, a little bit, somewhat, quite a bit, very much?"
* Ability to walk without requiring assistance from another individual (use of cane or walker acceptable)
* Normal organ and marrow function as defined below:

  * leukocytes >3,000/mcL
  * absolute neutrophil count >1,500/mcL
  * platelets >100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * creatinine clearance >30 mL/min
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Active malignancy or on-going cancer treatment including oral anti-estrogen therapy, immunotherapy, biologic therapy.
* Men receiving androgen deprivation therapy
* Use of Coumadin or Warfarin (other blood thinners are acceptable)
* Symptomatic congestive heart failure
* Lung disease requiring oxygen
* End stage renal disease requiring dialysis
* Inability to swallow capsules
* Chronic nausea or diarrhea defined by a frequency of ≥ once per week
* Hemoglobin <10 g/dl
* Diagnosis of dementia
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known untreated hypothyroidism
* Allergy to muscadine grapes or muscadine grape preparations

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Klepin, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klepin HD, Tooze JA, Bitting RL, Davis B, Pleasant K, Melo AC, Cook K, Soto-Pantoja DR, Tallant EA, Gallagher PE. Study design and methods for the pilot study of muscadine grape extract supplement to improve fatigue among older adult cancer survivors (FOCUS) trial. J Geriatr Oncol. 2023 May;14(4):101478. doi: 10.1016/j.jgo.2023.101478. Epub 2023 Mar 27. PMID 36990930

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm
Started | 32 | 32
Completed | 30 | 32
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.8 (5.4) | 75.8 (5.7) | 75.8 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 9 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 30 | 60
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 30 | 28 | 58
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Outcomes Measurement System (PROMIS) Fatigue 7a Questionnaire
Description: (PROMIS) Fatigue 7a will be used to assess fatigue. Using a mixed effects model with a constraint of a common baseline mean across treatment groups and an unstructured covariance matrix to model all fatigue measures over time, and use linear contrasts to estimate the difference in change and corresponding 90% confidence interval between the two groups. Item responses are rated on a five-point scale ranging from "never" to "always" and are summed for a total score and transformed to a T-score metric, which has a mean of 50 and a standard deviation of 10. Higher scores indicate more fatigue.
Time Frame: At baseline and at 12 weeks
Population: Not all participants reported data for this outcome measure.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm
Number analyzed (Participants) | 30 | 32
score on a scale | -6.6 (1.1) | -5.4 (2.2)
Statistical Analysis 1: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Test type: Superiority; Mean Difference (Final Values) = -1.2, 90% CI 2-sided [-3.5 to 1.1]

2. Secondary Outcome: Pepper Assessment Tool for Disability (PAT-D) Questionnaire - Change From Baseline at 12 Weeks
Description: Pepper Assessment Tool for Disability (PAT-D) will used to assess self-reported physical function. The (PAT-D) is a 19-item survey designed to assess domains of physical function in older adults which contains subscales on mobility, instrumental activities of daily living (IADLs), and basic activities of daily living (ADLs). Participant responses will best describe their ability to perform certain activities of daily living (On a scale of 1 to 5; 1 = usually did with no difficulty to 5 = unable to do. Minimum score of 19, max score of 95. A lower score indicates less difficulty with tasks and better function. Investigators will estimate 95% confidence intervals for the differences between the two groups for the secondary outcomes at 12 weeks reported as mean and standard error scores.
Time Frame: At 12 weeks
Population: Not all participants reported data for this outcome measure.
Measure: Mean (Standard Error); unit: mean score on a scale
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm
Number analyzed (Participants) | 29 | 30
mean score on a scale | 1.4 (0.1) | 1.6 (0.1)
Statistical Analysis 1: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Test type: Superiority; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]

3. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: The Short Physical Performance Battery (SPPB) will be used to objectively assess lower extremity physical function. This validated measure comprises a short walk, repeated chair stands, and balance test.
  Each section is scored out of 4 points, so the highest total score for the SPPB is 12 points. Score range is 0-12. Poor (0-6), moderate 7-9) and good (10-12). Lower scores on the SPPB have been associated with increased risk of disability, hospitalization and worse survival among older adults with and without cancer.
  Investigators will estimate 95% confidence intervals for the differences between the two groups for the secondary outcomes at 12 weeks.
Time Frame: At 12 weeks
Measure: Mean (Standard Error); unit: points
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm
Number analyzed (Participants) | 30 | 32
points | 9.8 (0.5) | 9.2 (0.5)
Statistical Analysis 1: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Test type: Superiority; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.7 to 2.0]

4. Secondary Outcome: Short Form Minnesota Leisure Time Activity Questionnaire (MLTA)
Description: This questionnaire will assess self-reported physical activity with participants answering yes/no questions in regards to physical activities done in the past two weeks and the frequency of those activities. Score is interpreted by calculating the total energy expenditure based on the frequency and duration of reported leisure activities, with higher scores indicating a greater level of physical activity; generally, scores are categorized as low (inactive), moderate (moderately active), and high (highly active). Investigators will estimate 95% confidence intervals for the differences between the two groups for the secondary outcomes at 12 weeks.
Time Frame: At 12 weeks
Measure: Mean (Standard Error); unit: kcal/week
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm
Number analyzed (Participants) | 30 | 32
kcal/week | 3218 (517) | 4192 (1141)
Statistical Analysis 1: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Test type: Superiority; Mean Difference (Final Values) = -973.5, 95% CI 2-sided [-3500 to 1553]

5. Secondary Outcome: 6-Minute Walk Test
Description: A 6-minute walk will be measured to assess physical fitness. The 6-minute walk is easy to administer in a clinical setting, accurately assesses submaximal exercise capacity, is an independent predictor of mortality and is correlated with peak V02 testing. The number of laps and distance walked on the final lap will be recorded. The total distance the participant walked will be entered onto the online database (1 lap = 30 meters distance). Investigators will estimate 95% confidence intervals for the differences between the two groups for the secondary outcomes at 12 weeks.
Time Frame: At 12 weeks
Population: Not all participants reported data for this outcome measure.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm
Number analyzed (Participants) | 29 | 29
meters | 369.8 (22.1) | 349.1 (14.4)
Statistical Analysis 1: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Test type: Superiority; Mean Difference (Final Values) = 20.7, 95% CI 2-sided [-32.4 to 73.8]

6. Secondary Outcome: Longitudinal Aging Study Amsterdam (LASA) Sedentary Behavior Questionnaire
Description: The questionnaire will be used to measure sedentary behavior for time spent during a 24 hour period for weekday and weekend various activities. The questionnaire consists of 10 items. The average time per 24 hours on each sedentary activity will be recorded in hours and/or minutes. Scores represent the self-reported average time an older adult spends engaged in sedentary activities (i.e., watching TV, reading, or sitting during a typical weekday and weekend day), with higher scores indicating a greater amount of time spent sedentary. Investigators will estimate 95% confidence intervals for the differences between the two groups for the secondary outcomes at 12 weeks.
Time Frame: At 12 weeks
Population: Not all participants reported data for this outcome measure.
Measure: Mean (Standard Error); unit: hours
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm
Number analyzed (Participants) | 30 | 32
hours | 13.2 (1.0) | 12.7 (0.9)
Statistical Analysis 1: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Test type: Superiority; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-2.2 to 3.2]

7. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Short Form (SF) - Quality of Life
Description: The PROMIS Global Health Short Form (SF) is a 10-item questionnaire that will assess global quality of life including overall physical health, mental health, social health, pain, fatigue an overall perceived quality of life. Participants will respond to questions or statements with varied selections (excellent to poor; completely to not at all; never to always; and none to very severe).
  Scores above 50 are considered a better than average quality of life and scores below 50 are considered below average quality of life.
  Higher T-scores indicate better health, so scores around 50 are average, while scores below 40 suggest poor health warranting further assessment, and scores above 60 indicate excellent health. 50 indicates the population mean with a standard deviation of 10 Investigators will estimate 95% confidence intervals for the differences between the two groups for the secondary outcomes at 12 weeks.
Time Frame: At 12 weeks
Population: Not all participants reported data for this outcome measure.
Measure: Mean (Standard Error); unit: T score
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm
Number analyzed (Participants) | 30 | 32
T score
  Quality of Life - Self-rate health | 3.4 (0.1) | 3.2 (0.1)
  Quality of life - Ability to carry out social activities and roles | 3.9 (0.2) | 3.7 (0.2)
  Physical health (t score) | 47.2 (1.2) | 46.3 (1.3)
  Mental health (t score) | 50.6 (1.5) | 52.0 (1.3)
Statistical Analysis 1: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Quality of Life - Self-rate health; Test type: Superiority; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.7]
Statistical Analysis 2: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Test type: Superiority — Quality of life - Ability to carry out social activities and roles; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.6]
Statistical Analysis 3: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Physical health (t score); Test type: Superiority; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-2.7 to 4.5]
Statistical Analysis 4: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Global Mental health (t score; Test type: Superiority; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.4 to 2.5]

8. Secondary Outcome: Adherence - Pill Count
Description: Adherence will be measured by pill count at study completion. Investigators will estimate 95% confidence intervals for the differences between the two groups for the secondary outcomes at 12 weeks.
Time Frame: 12 weeks
Population: Not all participants reported data for this outcome measure.
Measure: Mean (Standard Error); unit: number of pills
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm
Number analyzed (Participants) | 30 | 30
number of pills | 569.1 (35.4) | 568.0 (35.8)
Statistical Analysis 1: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Test type: Superiority; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-99.7 to 101.9]

9. Secondary Outcome: Fried Frailty Index
Description: Frailty indexes will be assessed for differences between the two arms. The Fried frailty index is a scoring system that classifies people into three stages of frailty based on five criteria: weight loss, exhaustion, low physical activity, and slowness. Frailty index scores can be calculated by dividing the sum of the recoded values of the variables by the number of variables measured for a person.
  Corresponding scores are: Score of 0, non-frail; score of 1-2 pre-frail; score of 3-5 frail. Higher scores represent higher rates of frailty among participants.
  Investigators will estimate 95% confidence intervals for the differences between the two groups for the secondary outcomes at 12 weeks.
Time Frame: At 12 weeks
Population: Not all participants reported data for this outcome measure.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm
Number analyzed (Participants) | 30 | 31
score on a scale | 0.9 (0.2) | 0.9 (0.2)
Statistical Analysis 1: Comparison: Muscadine Grape Extract Arm vs Placebo Arm; Test type: Superiority; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.5 to 0.5]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Muscadine Grape Extract Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/32
Other Adverse Events (participants affected / at risk) | 29/32 | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Muscadine Grape Extract Arm (N=32) | Placebo Arm (N=32)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Muscadine Grape Extract Arm (N=32) | Placebo Arm (N=32)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 6 (7)
Constipation (Gastrointestinal disorders) | 12 (13) | 9 (12)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 12 (14) | 12 (15)
Flatulence (Gastrointestinal disorders) | 12 (13) | 19 (22)
Nausea (Gastrointestinal disorders) | 4 (5) | 10 (11)
Fatigue (General disorders) | 4 (5) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT04495751/Prot_SAP_001.pdf
  • Informed Consent Form (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT04495751/ICF_000.pdf